CLINICAL TRIAL: NCT05324501
Title: Phase I Open Label Ascending Dose Study to Assess the Feasibility and Safety of Intermittent Infusions of MTX110 Administered by Convection-Enhanced Delivery (CED) in Patients With Recurrent Glioblastoma (rGBM) (MAGIC-G1)
Brief Title: A Study of Intra-tumoral Administered MTX110 in Patients With Recurrent Glioblastoma
Acronym: MAGIC-G1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Biodexa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MTX110-102
Record Dates: First submitted 2022-03-28; First posted 2022-04-12 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Two cohort 3+3 design. Between 4-18 patients per cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Cohort A: MTX-110 (Experimental): Weekly dosing of MTX110 via CED until progression/ unacceptable toxicity.
  Interventions: Drug: MTX110; Device: Programmable pump and catheter system
- Cohort B: MTX-110 with optional catheter repositioning (Experimental): Weekly dosing of MTX110 via CED until progression. At progression, optional catheter repositioning may occur, followed by continued weekly dosing of MTX110 until next progression/ unacceptable toxicity.
  Interventions: Drug: MTX110; Device: Programmable pump and catheter system

INTERVENTIONS:
Drug: MTX110 — Soluble panobinostat
Device: Programmable pump and catheter system — To allow Convection-Enhanced Delivery (CED)

SUMMARY:
A study designed to assess the safety of MTX110 in patients suffering with recurrent glioblastoma. MTX110 will be administered directly to the site of the tumour via a catheter which is inserted during a surgical procedure at the beginning of the study.

DETAILED DESCRIPTION:
A two cohort, ascending dose study of intra-tumoral MTX110 in patients with recurrent glioblastoma. With the aim to assess the safety and also the recommended phase 2 dose of MTX110.

The patient will undergo a surgical procedure to insert a programmable pump and catheter system to allow administration of MTX110 directly to the tumour using Convection Enhanced Delivery (CED).

Cohort A patients will receive one of three potential dose levels of MTX110 as a weekly infusion in order to establish recommended phase 2 dose. This will be based on an accelerated dose titration/3+3 design.

Cohort B patients will follow the 3+3 study design with the starting concentration established in Cohort A. They too will receive MTX110 as a weekly infusion and may undergo catheter repositioning and continued treatment following progression.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent glioblastoma.
* Patients must be healthy enough to tolerate surgery and general anesthesia.
* Estimated life expectancy of greater than 3 months.

Exclusion Criteria:

* Patients scheduled to undergo or are undergoing re-irradiation for the recurrent tumour.
* Patients with a history of glioblastoma treatment with carmustine or Gliadel® wafers.
* Patients who cannot undergo MRI.
* Patients may not have received chemotherapy or bevacizumab ≤ 4 weeks, or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week) prior to starting the study drug.
* Patients may not have received treatment with tumor treating fields ≤ 1 week prior to starting the study drug.
* Patients may not be less than 12 weeks from completion of radiation therapy for the primary tumor.
* Patients with neoplastic lesions in the brainstem, cerebellum, or spinal cord; radiological evidence of active; multifocal disease; extensive subependymal disease (tumor touching subependymal space is allowed); tumor crossing the midline or leptomeningeal disease.
* Posterior fossa location of the tumor, regardless of its morphology.
* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin (treatment with tamoxifen or aromatase inhibitors or other hormonal therapy that may be indicated in prevention of prior cancer disease recurrence, are not considered current active treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Safety of MTX110 administered by CED | Through study completion, an expected average of 28 weeks. DLT period 28 days from first dose.
  The frequency and nature of adverse events, serious adverse events and dose limiting toxicities (DLTs).
To determine the recommended Phase 2 dose (RP2D) of MTX110 | Through study completion, an expected average of 28 weeks

SECONDARY OUTCOMES:
Overall survival | 12 months
Progression-free survival | 6 months
  Progression based on mRANO criteria
Best overall response rate | 6 months
  Based on mRANO criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gary Shangold, Study Director — Biodexa Pharmaceuticals
Locations (2):
- United States (2):
  - Baptist MD Anderson, Jacksonville, Florida
  - Duke University Hospital, Durham, North Carolina